CLINICAL TRIAL: NCT02567526
Title: Cost Effectiveness of Nutrition Intervention in Long Term Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sandra Simmons, Associate Professor of Medicine, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 111645; 5R01AG033828 (NIH)
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Weight Loss
Keywords: food and fluid intake; nursing home residents; staffing
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care Control Group (No Intervention): Eligible, consented residents continued to receive usual care from nursing home staff and were monitored by trained research staff.
- Between-meal Intervention Group (Experimental): Non-nursing staff trained as Feeding Assistants were utilized to deliver supplements and snacks twice per day, between meals for 24 study weeks.
  Interventions: Behavioral: Between-Meal Intervention Group

INTERVENTIONS:
Behavioral: Between-Meal Intervention Group — Non-nursing staff trained as Feeding Assistants were responsible for supplement and snack delivery in the mornings and afternoons between meals supervised by research staff
  Arms: Between-meal Intervention Group

SUMMARY:
Inadequate food and fluid intake is a common problem among nursing home (NH) residents and one that can lead to under-nutrition, dehydration, weight loss, hospitalization, and even death. The most common nutrition intervention for at-risk NH residents is oral liquid nutrition supplementation, although, there is limited controlled evidence of the efficacy of supplements in promoting weight gain in NH residents. Moreover, studies show that supplements are not provided consistent with orders and residents receive little to no staff assistance to promote consumption in daily NH care practice. The result is that nutritionally at-risk NH residents with supplement orders receive few additional daily calories from supplements. Recent evidence strongly suggests that offering residents a choice among a variety of foods and fluids multiple times per day between meals coupled with assistance is effective in increasing daily caloric intake and promoting weight gain. However, the provision of the between-meal choice intervention requires significantly more staff time relative to the amount of time NH staff currently spend on between-meal nutritional care provision.

A new federal regulation allows NHs to train non-nursing staff to provide feeding assistance care. Preliminary research has demonstrated that non-nursing staff trained as "feeding assistants" provide mealtime feeding assistance care that is comparable to or better than their indigenous nurse aide counterparts. Moreover, a recent demonstration project showed that these staff can be used to effectively augment nurse aide staff for mealtime feeding assistance care provision in daily care practice. The proposed translational study will utilize the federal regulation to train non-nursing staff for between-meal nutritional care delivery. Specifically, the proposed study will use a controlled, intervention design to determine the cost-effectiveness of the between-meal choice intervention relative to a usual care control group in a group of 200 residents across 4 NH sites. Residents with an order for caloric supplementation will be included in this study and randomized into either a usual care control group or a choice intervention group (100 residents per group). The usual care control group will continue to receive standard NH care for supplement or snack delivery between meals, as provided by indigenous nurse aide staff. Non-nursing staff trained as "feeding assistants" will offer residents in the intervention group a choice between supplements and other snack foods and fluids twice daily, five days per week, for 24 weeks while also providing a standardized prompting protocol to enhance intake and independence in eating. Research staff will independently document the costs of intervention implementation and compare these costs to effectiveness measures which include improvements in caloric intake, weight and quality of life. These outcomes will be independently monitored for both groups across 24 study weeks by trained research staff using standardized, validated protocols. This translational research effort will provide critical information to improve care practices in nursing homes for nutritionally at risk residents.

ELIGIBILITY:
Inclusion Criteria:

* Long-stay nursing home residents
* Capable of oral food and fluid intake
* Physician or dietitian order for caloric supplementation

Exclusion Criteria:

* Short-stay (rehabilitation only)
* Feeding tube
* Hospice care
* History of Aspiration

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 148 (Actual)
Dates: Start 2011-08; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
total caloric intake during and between meals | 24 weeks
  Weighed intake methods were used to determine total caloric intake during and between meals before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sandra F Simmons, PhD, Principal Investigator — Vanderbilt University

REFERENCES:
- [Derived] Hollingsworth EK, Long EA, Simmons SF. Comparison Between Quality of Care Provided by Trained Feeding Assistants and Certified Nursing Assistants During Between-Meal Supplementation in Long-Term Care Settings. J Appl Gerontol. 2018 Nov;37(11):1391-1410. doi: 10.1177/0733464816669806. Epub 2016 Sep 22. PMID 27664171